CLINICAL TRIAL: NCT03139045
Title: Impact of VeinViewer® Vision to Guide Peripheral Venipuncture in Geriatrics
Acronym: VeinGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI2016_843_0030
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Venipuncture; Geriatric

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venous puncture using VVV at the beginning of the procedure (Active Comparator)
  Interventions: Biological: Venous puncture in elderly patients
- Venous puncture without VVV (Active Comparator)
  Interventions: Biological: Venous puncture in elderly patients

INTERVENTIONS:
Biological: Venous puncture in elderly patients — Venous puncture in elderly patients

SUMMARY:
Peripheral venipuncture is a common procedure in geriatrics. This procedure due to altered cutaneous alteration and venous capital associated with age poses problems of comfort and quality of life of elderly patients hospitalized. There is little data from the literature that highlights the difficulties of venipuncture in the context of old age. New venous visualization technologies by infrared spectroscopy (NIR) such as VeinViewer® Vision (VVV) have been developed to guide the placement of a peripheral venous (VVP) or venipuncture (PV) route.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 years and over
* Patient hospitalized in a department of acute geriatrics, whose venipuncture was prescribed

Exclusion Criteria:

* Patient not affiliated to a social security scheme
* Patient under legal protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Quantification of the number of attempts to place the venous catheter for venipuncture | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No